CLINICAL TRIAL: NCT06175390
Title: Tiragolumab, Atezolizumab and Chemotherapy in Triple Negative Breast Cancer: A Phase II Trial
Brief Title: Tiragolumab, Atezolizumab and Chemotherapy in Triple Negative Breast Cancer
Acronym: SKYLINE
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institut Curie (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IC 2022-01
Record Dates: First submitted 2023-11-27; First posted 2023-12-18 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Triple Negative Breast Cancer
Keywords: Triple Negative Breast Cancer; Atezolizumab; Tiragolumab; 68Ga-FAPI-46
MeSH Terms: conditions — Triple Negative Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: A phase II trial preceded by a safety run-in with two parallel cohorts
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort A: early Triple Negative Breast Cancer (Experimental): Patients will receive neoadjuvant therapy with four cycles of 1200 mg of atezolizumab and 600 mg of Tiragolumab every 3 weeks in combination with nab-paclitaxel 100 mg/m2 on days 1, 8, and 15, every 3 weeks plus carboplatin AUC 5 on days 1 every 3 weeks then four cycles of 1200 mg of atezolizumab (Tecentriq®, Roche) and 600 mg of Tiragolumab (Roche) every 3 weeks in combination with Doxorubicin 60 mg/m2 plus Cyclophosphamide 600 mg/m2.
  After surgery, patients will receive adjuvant treatment with atezolizumab plus tiragolumab every 3 weeks for up to nine cycles (in patients with germline BRCA1/2 mutation eligible to adjuvant olaparib, tiragolumab and atezolizumab will not be resumed after surgery).
  Interventions: Radiation: 68Ga-FAPI-46 PET/CT; Biological: Tumor samples analysis; Biological: Blood samples analysis: Circulating Tumor DNA
- Cohort B: metastatic Triple Negative Breast Cancer (Experimental): Patients will receive atezolizumab 1680 mg administered by IV infusion Q4W, plus tiragolumab 840 mg administered by IV infusion Q4W, plus nab-paclitaxel 100 mg/m2 administered by IV infusion d1, d8, d15 of every 28-day cycle.
  Treatments will be administered until disease progression or limiting toxicity.
  Interventions: Radiation: 68Ga-FAPI-46 PET/CT; Biological: Tumor samples analysis; Biological: Blood samples analysis: Circulating Tumor DNA

INTERVENTIONS:
Radiation: 68Ga-FAPI-46 PET/CT — Cohort A:
  Tumor assessments by 18F-FDG PET/CT (per PERCIST v1.0) will be performed at: baseline, after the first 2 treatment cycles (between C2D15 and C3D1), and before surgery (after the last administration of neoadjuvant chemotherapy) Tumor assessment by 68Ga-FAPI-46 PET/CT will be performed at: baseline and before surgery (after the last administration of neoadjuvant chemotherapy).
  Cohort B:
  Tumor assessments by 18F-FDG PET/CT per PERCIST v1.0 will be performed at baseline, every 8 weeks (+/- 1 week) for the first 24 weeks, and every 12 weeks (+/- 1 week) thereafter until disease progression or treatment discontinuation, whichever is later.
  Tumor assessments by 68Ga-FAPI-46 PET/CT will be performed at baseline and after the first 2 treatment cycles and will be synchronized with 18F-FDG PET/CT.
Biological: Tumor samples analysis — Patients will undergo a mandatory biopsy of the primary tumor at baseline, after the first 2 treatment cycles and during the surgery. A lymph node biopsy will be performed at baseline if feasible in cohort A, and and in case of disease progression for cohort B (if clinically feasible).
  In addition to the usual morphological and immunohistochemical (ER, PR, HER2+, CPS score, PD-L1 status with SP142 …) analyses in the cohort A and cohort B , exploratory analyses will be performed.
Biological: Blood samples analysis: Circulating Tumor DNA — Blood samples will be collected at baseline. In addition for cohort A at cycles 2 and 3, within 21 days before surgery, 10 to 21 days after surgery and at cycle 8 after surgery. In addition for cohort B after the first 2 treatment cycles and in case of disease progression (if clinically feasible).

SUMMARY:
This is a phase II study, preceded by a safety run-in, with two independent cohorts (cohort A in early Triple Negative Breast Cancer (TNBC) patients and cohort B in late in metastatic TNBC patients) designed to evaluate the efficacy of atezolizumab, tiragolumab and chemotherapy.

DETAILED DESCRIPTION:
In the early TNBC setting (cohort A) dedicated to patients with newly diagnosed, previously untreated, non-metastatic disease (tumor stage T1c, nodal stage N1-2, or tumor stage T2-4, nodal stage N0-2), the treatment will consist in:

First part: Nab-paclitaxel administered weekly in combination with atezolizumab, tiragolumab and carboplatin, administered every 3 weeks over 12 weeks Second part: Atezolizumab, tiragolumab, doxorubicin and cyclophosphamide, administered every 3 weeks over 12 weeks Patients will undergo surgery of the primary disease 3 to 6 weeks after last neoadjuvant treatment dose, followed by 9 cycles of atezolizumab and tiragolumab administered every 3 weeks.

Treatment efficacy will be assessed early on, through 18F-FDG PET/CT during the first two cycles. Patients whose tumor shows no sign of response after two cycles (i.e. no partial or complete metabolic response of the breast tumor according to 18F-FDG PET/CT by PERCIST criteria) would then be switched to standard treatment, per investigator decision.

Tiragolumab 600 mg and Atezolizumab 1200 mg administered by IV infusion every 3 weeks after surgery for a total of 9 cycles.

In the metastatic TNBC setting (cohort B) dedicated to patients with locally recurrent inoperable or metastatic disease eligible to first line treatment, patients will be included regardless of their PD-L1 tumor expression defined by immunohistochemistry (Ventana SP142) at baseline, but no more than 40% of PD-L1 negative (i.e <1%) will be included. The treatment will consist in nab-paclitaxel administered at d1, d8, d15 of every 28-day cycle, combined with atezolizumab and tiragolumab administered every 3 weeks until disease progression or limiting toxicity.

Treatments will be administered until disease progression or limiting toxicity.

As the the combination Atezolizumab + Tiragolumab + chemotherapy has never been tested, a safety run-in phase of 10 patients is planned in each cohort to verify the tolerance of the combination

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old
2. Female
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
4. Histological diagnosis of carcinoma of the breast, according to AJCC 8th edition that is estrogen receptor negative (ER-), progesterone receptor negative (PR-) and HER2- negative according to local testing on the most recent tumor sample examined before signing consent form to participate in the study.

   1. ER-negative and PR-negative are defined as having an immunohistochemistry (IHC) < 10%
   2. HER2 negative is defined as per the 2018 American Society of Clinical Oncology (ASCO) - College of American Pathologists (CAP) guidelines, indeed as having an IHC of 0 or 1+ without ISH OR IHC 2+ and ISH non-amplified with ratio less than 2.0 and if reported, average HER2 copy number < 4 signals/cells OR ISH non-amplified with ratio less than 2.0 and if reported, average HER2 copy number < 4 signals/cells [without IHC]; Note: a IHC of 3+ is always considered HER2 positive, independently of the ISH result.

   Cohort A (early setting): patients will be enrolled regardless of their tumor PD-L1 status.

   Cohort B (metastatic setting): patients will be enrolled regardless of their tumor PD-L1 status but participants with PD-L1 negative tumor status (i.e.<1% defined by Immunohistochemistry with Ventana SP142) will be capped at 40%. i.e.<1% defined by immunohistochemistry with Ventana SP142) will be capped at 40%.
5. Agreement to perform new study-related biopsies and blood sampling as described in the study schedule of activity.
6. Tumor considered as accessible by biopsy, according to the investigator. Fine-needle aspiration, brushing, cell pellet from pleural effusion, bone metastases, and lavage samples are not acceptable. Tumor tissue from bone metastases is not acceptable.
7. For female of childbearing potential (WCBP): negative serum or urinary pregnancy test within 2 weeks prior to first dose of study administration.
8. Women of childbearing potential must agree to use one highly effective method of contraception during the screening period, during the course of the study and at least 12 months after the last administration of study treatment (see appendix 7) .
9. Adequate bone marrow function as defined below:

   Absolute neutrophil count ≥1500/μL, i.e., 1.5x109/L Hemoglobin ≥ 9.0 g/dL Platelets ≥100000/μL, i.e., 100x109/L
10. Adequate liver function as defined below:

    Serum total bilirubin ≤ 1.5 x ULN. In case of known Gilbert's syndrome ≤ 3 x UNL is allowed AST ≤ 3.0 x ULN, ALT ≤ 3.0 x ULN
11. Adequate renal function as defined below:

    Creatinine ≤ 1.5 x UNL and eGFR≥40ml/min/1.73m²
12. Adequate coagulant function as defined below:

    International Normalized Ratio (INR) ≤ 1.5 x ULN
13. Completion of all necessary screening procedures within 28 days prior to inclusion
14. Signed Informed Consent form (ICF) obtained prior to any study related procedure
15. Patients must be covered by a health insurance system

    Inclusion criteria #16 to #18 are applicable to cohort A (early setting):
16. For tumor stage T1c, nodal stage N1-3, by at least one radiographic or clinical measurement.

    For tumor stage T2-4, nodal stage N0-3, by at least one radiographic or clinical measurement.
17. Multifocal, multicentric unilateral or bilateral breast adenocarcinoma tumors are allowed provided that all foci are ER-/PR-/HER2- according to local testing.
18. Left ventricular ejection fraction (LVEF) ≥ 50%.

    Inclusion criteria #19 to 23 are applicable to cohort B (metastatic setting):
19. No prior line of chemotherapy / or systemic therapy for metastatic disease (patients with known germline BRCA1 or BRCA2 mutations may have been treated with one prior line of therapy with PARP inhibitor).
20. Radiation therapy for metastatic disease is permitted. There is no required washout period for radiation therapy. Patients should be recovered from the effects of radiation.
21. Prior chemotherapy in the neoadjuvant or adjuvant setting is allowable if treatment was completed 12 months prior to inclusion.
22. Patients with documented liver metastases: AST and ALT Patients with documented liver metastases: AST and ALT less than 5 x ULN
23. Have a life expectancy of at least 3 months.

Exclusion Criteria:

1. Pregnant and/or lactating women.
2. Contra-indications to 18F-FDG PET/CT and/or 68Ga-FAPI-46 PET/CT.
3. Patients in whom tumor deposits are not detected by 18F-FDG PET/CT.
4. Subject with a significant medical, neuro-psychiatric, substance abuse or surgical condition, currently uncontrolled by treatment, which, in the principal investigator's opinion, may interfere with completion of the study.
5. TNM stage T4d breast cancer (inflammatory breast cancer).
6. Known HIV
7. Active infection including: Hepatitis B (known positive HBV surface antigen (HBsAg) result). Subjects with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible; Hepatitis C. Subjects positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
8. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, active tuberculosis, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the subject to give written informed consent.
9. Concomitant use of other investigational drugs.
10. Any unresolved toxicity NCI CTCAE Grade ≥2 from previous anticancer therapy with the exception of alopecia. Subjects with Grade ≥2 neuropathy will be evaluated on a case-by-case basis after consultation with the Study Physician.
11. Active or prior documented autoimmune disease (including inflammatory bowel disease, celiac disease, Wegener's granulomatosis) within the past 3 years.

    Note: Subjects with childhood atopy or asthma, vitiligo, alopecia, Grave's disease, Hashimoto's thyroiditis, on a stable dose of thyroid replacement hormone or psoriasis not requiring systemic treatment (within the past 2 years), and patients with controlled Type 1 diabetes mellitus on a stable insulin regimen are not excluded.
12. Known history of, or any evidence of active, non-infectious pneumonitis. (Note: History of radiation pneumonitis in the radiation field [fibrosis] is permitted).
13. History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins.
14. Known hypersensitivity or allergy to biopharmaceuticals produced in Chinese hamster ovary (CHO) cells or any component of the atezolizumab formulation.
15. Any live (attenuated) vaccine within 30 days of planned start of study therapy.
16. Treatment with systemic immunosuppressive medications (including but not limited to corticosteroids, cyclophosphamide, azathioprine, cyclosporine, methotrexate, thalidomide, and antitumor necrosis factor [TNF] agents) within 2 weeks prior to inclusion, or anticipated requirement for systemic immunosuppressive medications during the trial.

    1. Patients who have received acute, low-dose (≤ 10 mg oral prednisone or equivalent), systemic immunosuppressant medications may be enrolled in the study.
    2. The use of corticosteroids (≤10 mg oral prednisone or equivalent) for chronic obstructive pulmonary disease, mineralocorticoids (e.g., fludrocortisone) for patients with orthostatic hypotension, and low dose supplemental corticosteroids for adrenocortical insufficiency are allowed.
17. Prior treatment with anti-PD-1 or anti-PD-L1 therapeutic antibody within 6 months.
18. Prior allogeneic stem cell or solid organ transplantation
19. Known active EBV
20. Known lymphoepithelioma-like carcinoma
21. Patients with an obstruction of urine flow (according to the current SmPc of cyclophosphamide)
22. Oligometastatic patients if they require locoregional treatment.

    Exclusion criteria #23 to #25 are applicable to cohort A (early setting):
23. Presence of any distant metastasis.
24. Known germline BRCA1 or BRCA2 mutation.
25. Contra-indication for treatment by nab-paclitaxel, doxorubicin, cyclophosphamide, carboplatin or known allergy to any tested substances or any excipients (e.g; chemotherapy or immunotherapy formulations).

    Exclusion criteria #26 to #28 are applicable to cohort B (metastatic setting):
26. Contra-indication for treatment by nab-paclitaxel or known allergy to any tested substances or any excipients (e.g; chemotherapy or immunotherapy formulations).
27. Leptomeningeal disease and known CNS disease, except for treated asymptomatic CNS metastases, provided all of the following criteria are met:

    Only supratentorial and cerebellar metastases allowed (i.e., no metastases to midbrain, pons, medulla, or spinal cord) Treated and stable CNS metastases since at least 4 weeks before inclusion No ongoing requirement for corticosteroids as therapy for CNS disease No stereotactic radiation within 7 days or whole brain radiation within 14 days prior to inclusion No evidence of interim progression between the completion of CNS-directed therapy and the screening radiographic study Note: asymptomatic brain metastases discovered during the screening, by e.g. 68Ga-FAPI-46 PET/CT and deemed accessible to stereotactic radiation therapy could remain in the study after discussion with the study medical monitors.
28. Prior malignancy other than breast cancer active within the previous 5 years, except for localized cancers that are considered to have been cured and in the opinion of the investigator present a low risk for recurrence. Examples include basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the cervix or breast.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2024-03-27 (Actual); Primary Completion 2026-08-15 (Estimated); Study Completion 2029-02-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability]. | 6 weeks for cohort A and 8 weeks for cohort B
  In Safety run-in, safety and toxicity of the combination Atezolizumab + Tiragolumab + chemotherapy in cohorts A
In cohort A, Rate of pathological complete response (pCR) | 6 months
  pCR is defined as ypT0/Tis ypN0 (i.e., no invasive residual in breast or nodes; as centrally assessed at the time of definitive surgery).
In cohort B, Progression-free survival rate (6mPFS), | 6 months
  6mPFS is defined as the proportion of patients without progression (as assessed by central review per Positron Emission Tomography Response Evaluation Criteria in Solid Tumors (PERCIST) v1.0) or death within 6 months after the date of inclusion.

SECONDARY OUTCOMES:
SAEs (serious adverse events) and AEs (adverse events) | 36 months
  SAEs and AEs will be assessed according to NCI CTCAE v5.0, by grade and their relationship to atezolizumab and/or tiragolumab and/or chemotherapy.
In Cohort A, alternative definition of pCR rate: Residual cancer burden (RCB) | 6 months
  Residual cancer burden (RCB) classes according to the MD Anderson classification as assessed per central assessment.
In Cohort A, alternative definition of pCR rate: ypT0 ypN0 (no invasive or noninvasive residual in breast or nodes | 6 months
  ypT0 ypN0 defined per central assessment.
In Cohort A, Invasive disease-free survival (iDFS) | 3 years
  3 years-iDFS defined as the time from inclusion to occurrence of any of the following: ipsilateral invasive breast cancer recurrence, regional invasive breast cancer recurrence, distant recurrence, death attributable to any cause, contralateral invasive breast cancer, or second non-breast invasive cancer, whichever comes first.
In Cohort B, Objective response rate (ORR) | 6 months
  ORR defined as the proportion of patients who have a complete response (CR) or partial response (PR) based on local investigator assessment, per PERCIST 1.0 among patients with measurable disease at baseline.
In Cohort B, Duration of response (DoR) | 3 years
  DoR defined as the time from the date of first documented response until date of documented progression per PERCIST 1.0 based on local investigator assessment or death due to any cause.
In Cohort B, Clinical benefit rate (CBR) | 6 months
  6-month-CBR defined as the proportion of patients who have achieved either a confirmed complete or partial response, or stable disease for at least 24 weeks after treatment start per PERCIST 1.0 based on local investigator assessment.
Quality of Life mesurement with 5 Dimension 5 Level scale Questionnaire | 6 months
  The scale measures quality of life on a 5-component scale including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The five states in the EQ-5D-5L are referred to by 5-digits, score from 11111 to 55555. Each number is added up to produce a score between 5 and 25 for EQ-5D-5L.
Overall Survival (OR) | 5 years
  OS defined as the time from inclusion to the date of death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: François-Clément Bidard, PhD, Principal Investigator — Institut Curie
Locations (2):
- France (2):
  - Institut Curie, Paris
  - Institut Curie, Saint-Cloud

IPD SHARING:
Plan to Share IPD: Yes
Sponsor will share de-identified data sets. Documents generated under the project will be disseminated in accordance with Institut Curie policies.
Supporting Information: Study Protocol, SAP
Time Frame: Data requests can be submitted starting 9 months after last article publication and will be made accessible for up to 12 months.
Access Criteria: Access to trial individual participant data can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a data sharing agreement (DSA).